CLINICAL TRIAL: NCT06160934
Title: The T1D Parent Check-In: A Preventative Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ellen H. O'Donnell, Assistant Professor Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023P002600
Record Dates: First submitted 2023-11-20; First posted 2023-12-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes; Diabetes in Children
Keywords: Pediatrics; Pediatric Endocrinology; Parenting Intervention; Pediatric Type 1 Diabetes; Pediatric Psychology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups: the T1D Parent Check-in Intervention group or the Treatment as Usual Group (TAU). Participants in the intervention and TAU groups will be yoked by age group (e.g., parent of an 8-12-year-old child will be yoked to another parent of an 8-12-year-old child) to minimize variability in effects due to differences in parenting by child age. Matching participants by clinic location (e.g., child receiving care at MGH will be yoked to another child receiving care at MGH) will serve as a natural control for differences in practice between clinic locations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The T1D Parent Check-in Group (Intervention Group) will participate in three sessions that will be delivered by a licensed clinical psychologist. In the larger RCT, the intervention will be manualized with training and a treatment protocol that can be delivered by any trained member of the diabetes psychosocial team (e.g., social workers, licensed mental health clinicians, and/or clinical psychologists). The intervention is designed to be both tailored and flexible but with fidelity to a basic structure. Diabetes-specific handouts and videos will be created as part of the intervention and will be provided to families throughout the course of the study.
  Interventions: Behavioral: T1D Parent Check-in
- Treatment as Usual (TAU) Group (No Intervention): Parents assigned to the Treatment As Usual (TAU) group will complete T1-T4 study questionnaires alongside the intervention group. They will also take the Motivation Quiz as part of their T2 questionnaires. Instead of a one-month phone call, these participants will be scheduled for a one-time consultation with a study psychologist after completing their T4 questionnaires. This consultation will entail reviewing the family's specific questionnaire results, discussing challenges/strategies relevant to the family's needs, and providing additional recommendations/referrals as indicated. Families will also be provided access to study resources that will assist with their family's overall adjustment to T1D.

INTERVENTIONS:
Behavioral: T1D Parent Check-in — The Type 1 Diabetes (T1D) Parent Check-in is an innovative, 3-session, T1D-specific intervention for parents of newly diagnosed children and adolescents that can be delivered via telehealth. The T1D Parent Check-in is an adaptation of The Parent Check-In, a brief, prevention-based parenting intervention developed by Grolnick, Levitt, Caruso, & Lerner (2021). The T1D Parent Check-in is designed to promote parenting skills on dimensions of autonomy support, structure and involvement that facilitate children's adjustment and motivation, and integrates skills from cognitive-behavioral therapy, customized to be highly relevant to families with a child 6-12 months from new diagnosis of T1D. The intervention is intended to promote diabetes-related resilience and positive psychological and medical outcomes among families of children with T1D.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn how to best support families during the first year of a child or teen's Type 1 diabetes (T1D) diagnosis. Specifically, we are testing a parenting intervention, the T1D Parent Check-in, designed for parents of children, ages 8 to 17 years, who have been newly diagnosed with T1D. This three-session intervention is delivered by diabetes psychologists over telehealth with the goal of helping families adjust to T1D, build resilience, and improve children's long-term health.

For this trial, our main question is whether parents like the intervention and find it to be helpful and worth their time and effort. We also want to test whether participating in the intervention helps parents feel more confident in their parenting and problem-solving around diabetes, feel less worried about diabetes, reduce family conflict, and improve children's quality of life. To answer these questions, we will randomly assign study participants to one of two groups; parents will either 1) receive the T1D Parent Check-in intervention, or 2) receive their usual care through clinic. Parents assigned to the second group will have the option of participating in a one-time meeting with the psychologist at the end of the study to receive general information/resources from the study and receive feedback on their questionnaires. Parents in both groups will be asked to complete questionnaires four times over the course of six months. Parents will be paid to complete the questionnaires.

DETAILED DESCRIPTION:
The purpose of the project is to develop and pilot an innovative, 3-session, Type 1 Diabetes-specific telehealth intervention for parents of newly diagnosed children and adolescents. This study is a multi-method, mixed quantitative and qualitative pilot project that will inform a future randomized control trial (RCT). The intervention will be piloted at two pediatric diabetes clinics: Massachusetts General Hospital (MGH) for Children and Boston Children's Hospital (BCH). Families of patients ages 8-17 years diagnosed with T1D within the past 3-9 months will be invited to participate in the study and then be randomly assigned to either the intervention group or a treatment-as-usual (TAU) group, with a goal of 25 families per group.

Measures of key outcomes (i.e., feasibility and acceptability measures, measures of diabetes-related resilience, distress, and family conflict, problem-solving, parenting style, parental stress, parent/child adjustment to children's chronic illness diagnosis, and health mindsets) will be collected via parent survey at baseline (T1), post-intervention (T2), 1-month follow-up (T3) and 6-month follow-up (T4) for within and between groups analyses. Qualitative feedback on the intervention will be sought from participating families after the third session (T2) and feedback on families' needs in the first year of diagnosis will be sought from all participants at T4. Additional information will be gathered from the medical record on diabetes regimen, HbA1c and demographics for descriptive statistics. This will also allow for exploratory analysis of change in HbA1c pre- to post-intervention and differences in glycemic control between groups.

ELIGIBILITY:
Inclusion Criteria:

* Parents/ primary caregivers (aged >18) of pediatric patients (ages 8-17 years), who have been diagnosed with T1D for at least 3 months, but not greater than 9 months (to ensure the intervention can be delivered within the first year of diagnosis)
* At least one caregiver (>18) proficient in the English language, as neither the intervention nor scales used in the study have been validated in other languages. The age range of the patient with diabetes 8-17 was chosen to include both middle childhood and adolescence when diagnosis of Type 1 diabetes is most common.

Exclusion Criteria:

* Parents' developmental delay or other cognitive impairment that may interfere with their completion of questionnaires or understanding of psychoeducational concepts, and
* Parental scores in the "severe" range of depression and anxiety, evaluated using routine screening measures for depression and anxiety and which may indicate the parent requires a higher level of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, an average of 8 months
  Recruitment data measured by percent of eligible families that were approached for participation that enrolled in study.
Intervention Completion Rate | Through study completion, an average of 8 months
  Feasibility of the intervention measured by percentage of intervention group participants who complete all three sessions of the intervention.
Client Satisfaction Questionnaire | Through study completion, an average of 8 months
  Participants in the intervention arm will complete the standardized Client Satisfaction Questionnaire (CSQ), a measure of overall satisfaction with the intervention.

SECONDARY OUTCOMES:
Parenting in Pediatric Diabetes Questionnaire | Through study completion, an average of 8 months
  Parents will rate their parenting in relation to their children's diabetes management.
Health Mindset Scale | Through study completion, an average of 8 months
  Parents will complete the Health Mindset Scale, rating their beliefs about health as more changeable versus fixed.
Diabetes Problem Solving Interview (DPSI) | Through study completion, an average of 8 months
  Parents will complete the standardized DPSI interview to evaluate diabetes-specific problem-solving.
Parent Problem Areas in Diabetes for Children and Teens | Through study completion, an average of 8 months
  Parents will complete the standardized Parent Problem Areas in Diabetes for Children and Teens to evaluate diabetes-related distress.
Diabetes Family Conflict Scale | Through study completion, an average of 8 months
  Parents will complete the Diabetes Family Conflict Scale - Parent Report (DFCS) and rate how often they argued with their children over the past month across various tasks of diabetes management (e.g., remembering to check blood sugars).
Connor-Davidson's Resilience Scale (CD-RISC-10) | Through study completion, an average of 8 months
  Parents will complete the Connor-Davidson's Resilience Scale (CD-RISC-10), a widely used measure of psychological resilience.
Parenting Efficacy | Through study completion, an average of 8 months
  The Parenting Efficacy scale measures parents' perceptions of efficacy in their parenting role.
Type 1 Diabetes and Life (T1DAL) | Through study completion, an average of 8 months
  Parents will reflect on their own quality of life as a parent of a child or teen with T1D by completing the standardized Type 1 Diabetes and Life (T1DAL) measure.
Child Hemoglobin A1C | Through study completion, an average of 8 months
  The child's most proximate HbA1C value will be collected from their electronic medical record.
Time in Range | Through study completion, an average of 8 months
  Children's prior one month time in range (TIR) will be collected for patients on continuous glucose monitors (CGM).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No